CLINICAL TRIAL: NCT07246434
Title: Efficacy of Platelet-Rich Plasma Versus Home-Based Exercise in Patients With Partial-Thickness Supraspinatus Tears: A Prospective Controlled Study
Brief Title: Platelet-Rich Plasma Versus Home-Based Exercise for Partial-Thickness Supraspinatus Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carlos Fernández-Morales, Clinical Professor, Universidad de Extremadura
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Rotator Cuff Injuries; Shoulder Joint; Shoulder Pain
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Two-group prospective controlled design comparing PRP injections with a home-based exercise program in parallel arms.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP Injection (Experimental): Participants receive three monthly ultrasound-guided intratendinous injections of platelet-rich plasma (PRP) in the affected supraspinatus tendon, preceded by local anesthetic infiltration in the subacromial bursa.
  Interventions: Biological: Platelet-Rich Plasma (PRP)
- Home-Based Exercise Program (Active Comparator): Active Comparator
  Interventions: Other: Home Exercise Program

INTERVENTIONS:
Biological: Platelet-Rich Plasma (PRP) — Ultrasound-guided intratendinous injection of 4 mL PRP prepared from autologous blood using the BS PRP SYSTEM-20 kit. A total of three injections are administered at one-month intervals. Local anesthesia with 5 mL mepivacaine 2% is applied subacromially prior to PRP administration.
  Arms: PRP Injection
Other: Home Exercise Program — A supervised-prescribed home-based shoulder exercise program including mobility, strengthening, and scapular stabilization exercises. The program is performed regularly over approximately three months, with progression based on clinical guidelines for rotator cuff rehabilitation.
  Arms: Home-Based Exercise Program

SUMMARY:
This study evaluates the clinical effectiveness of platelet-rich plasma (PRP) injections compared with a home-based exercise program in patients with partial-thickness tears of the supraspinatus tendon. Partial supraspinatus tears are a common cause of chronic shoulder pain and functional limitation. PRP has been proposed as a biological treatment that may promote tissue healing, while therapeutic exercise remains a standard conservative intervention.

This prospective, controlled study includes two parallel groups. The PRP group receives three monthly ultrasound-guided intratendinous PRP injections, preceded by local anesthesia. The control group follows a structured home-based exercise program for the same overall treatment period. All participants are assessed at baseline and again two months after completing their assigned intervention.

The primary outcome is shoulder pain measured with a Visual Analog Scale (VAS). Secondary outcomes include shoulder range of motion (flexion, extension, abduction, adduction, internal and external rotation) and functional disability measured with the Constant-Murley Score. The study also analyzes whether patient characteristics such as age or sex are associated with clinical improvement.

The aim of this research is to compare two commonly used conservative treatment strategies and provide evidence to guide clinical decision-making for patients with partial-thickness supraspinatus tears.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 70 years.

Shoulder pain for more than 6 months with a Visual Analog Scale (VAS) score > 4.

Partial-thickness tear of the supraspinatus tendon confirmed by ultrasound.

No improvement in VAS after conservative treatment with NSAIDs and/or physical therapy during the previous 6 months.

Willingness to undergo blood extraction and PRP infiltrations as required by the protocol.

Exclusion Criteria:

* Age < 20 or > 70 years.

Full-thickness tear of the supraspinatus tendon.

Active infection (osteomyelitis, septic arthritis).

Current treatment with NSAIDs, antiplatelet agents, or systemic immunosuppressants.

Severe thrombocytopenia.

Positive serology (syphilis, HIV, HBV, HCV).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain (VAS) | Baseline and 2 months after completing the intervention.
  Pain intensity measured using a 0-10 Visual Analog Scale (VAS). Higher scores indicate greater pain.

SECONDARY OUTCOMES:
Shoulder Range of Motion (Flexion, Extension, Abduction, Adduction, Internal and External Rotation) | Baseline and 2 months after completing the intervention.
  Active shoulder range of motion measured using standard goniometry in degrees.
Constant-Murley Score | Baseline and 2 months post-intervention.
  Composite functional score assessing pain, daily activities, range of motion, and strength. Total score ranges from 0 to 100; higher scores indicate better shoulder function.
Roles and Maudsley Score | Baseline and 2 months post-intervention.
  Four-point scale evaluating patient-perceived outcome (1 = excellent, 4 = poor).
QuickDASH Score | Baseline and 2 months post-intervention.
  Disability and symptoms of the upper limb measured with the QuickDASH questionnaire (0-100 scale). Higher scores indicate greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo-Antúnez, Ph.D., Study Director — University of Extremadura
Locations (1):
- University of Extremadura, Badajoz, Badajoz, Spain